CLINICAL TRIAL: NCT00029107
Title: Rituximab (Anti-CD20) for the Treatment of Hepatitis C Associated Cryoglobulinemic Vasculitis
Brief Title: Rituximab to Treat Hepatitis C-Associated Cryoglobulinemic Vasculitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Michael C Sneller, MD, Medical Officer, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 020096; 02-I-0096 (Other: NIAID Intramural protocol number)
Record Dates: First submitted 2002-01-05; First posted 2002-01-07 (Estimated); Results first posted 2012-04-03 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-04

CONDITIONS: Hepatitis C; Vasculitis
Keywords: Hepatitis; Vasculitis; Rituximab; Cryoglobulinemia; Hepatitis C; HcV-cV; Cryoglobulinemic Vasculitis
MeSH Terms: conditions — Hepatitis C; Vasculitis; Hepatitis; Cryoglobulinemia; Cryoglobulinemia, Familial Mixed | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate treatment (Other): Patients receive treatment with four weekly infusions of rituximab 375mg/m2 immediately following randomization.
  Interventions: Drug: Rituximab
- Delayed treatment (Other): Patients treated with standard therapy (corticosteroids, plasma exchange, etc.). After 6 months, they are eligibile to cross over and receive four weekly infusions of rituximab.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — anti-CD20 monoclonal antibody

SUMMARY:
The purpose of this study is to assess the efficacy of Rituximab (anti-CD20) in the treatment of patients with hepatitis C associated cryoglobulinemic vasculitis (HCV-CV) who have failed or are intolerant to interferon-alpha/ribavirin therapy. Up to 75 patients may be screened to enroll 34 adult patients with active HCV-CV in this randomized, non-blinded phase I/II trial. Patients will be randomized to receive either Rituximab 375 mg/M(2) on days 1, 8, 15 and 22 beginning at the time of enrollment or standard therapy. Patients in both groups will be maintained on stable doses of any immunosuppressive therapies that they were receiving at the time of enrollment. Response to Rituximab will be assessed by clinical and laboratory parameters.

Although the cause of cryoglobulinemic vasculitis is not known, a critical component is the presence of cryoglobulins-abnormal proteins that white blood cells called B lymphocytes produce in response to the chronic hepatitis C infection. Rituximab decreases the number of B cells. The Food and Drug Administration approved Rituximab in 1997 for the treatment of B-cell non-Hodgkin's lymphoma.

Patients between 18 and 75 years of age with hepatitis C and signs and symptoms of cryoglobulinemic vasculitis may be eligible for this study. They must have failed, or been unable to tolerate, treatment with IFN-a and ribavirin. Candidates will be screened with a history and physical examination, electrocardiogram (ECG), blood and urine tests, 24-hour urine collection and chest X-ray, if clinically indicated.

Participants will be randomly assigned to receive Rituximab upon entering the study or 6 months after entering the study. Those whose treatment is delayed 6 months will be followed once a month at NIH for disease evaluation and blood tests during that time.

Patients will be given Rituximab intravenously (through a vein) once a week for 4 weeks. For the first dose, patients will be admitted to the hospital for at least 24 hours after the infusion for monitoring. Subsequent infusions will be given on an inpatient or outpatient basis, depending on how the infusion is tolerated. The day before each infusion they will have a history and physical examination, blood work, and other tests, such as X-rays, as clinically indicated.

After the four infusions, patients will be followed for drug side effects and response to treatment. They will have blood tests every week for 4 weeks and will then return to NIH for 1 day every month for 12 months for a physical examination, blood tests, and X-rays, if medically indicated. Visits may be more frequent, if necessary, and patients may be asked to stay longer than a day if test findings requ...

DETAILED DESCRIPTION:
Although the cause of cryoglobulinemic vasculitis is not known, a critical component is the presence of cryoglobulins-abnormal proteins that white blood cells called B lymphocytes produce in response to the chronic hepatitis C infection. Rituximab decreases the number of B cells. The Food and Drug Administration approved Rituximab in 1997 for the treatment of B-cell non-Hodgkin's lymphoma.

Patients between 18 and 75 years of age with hepatitis C and signs and symptoms of cryoglobulinemic vasculitis may be eligible for this study. They must have failed, or been unable to tolerate, treatment with IFN-a and ribavirin. Candidates will be screened with a history and physical examination, electrocardiogram (ECG), blood and urine tests, 24-hour urine collection and chest X-ray, if clinically indicated.

Participants will be randomly assigned to receive Rituximab or standard therapy for 6 months after entering the study. All patients will be followed once a month at NIH for disease evaluation and blood tests during that time.

Patients will be given Rituximab 375 mg/m2intravenously once a week for 4 weeks. The day before each infusion they will have a history and physical examination, blood work, and other tests, such as X-rays, as clinically indicated.

After the four infusions, patients will be followed for drug side effects and response to treatment. They will have blood tests every week for 4 weeks and will then return to NIH for 1 day every month for 12 months for a physical examination, blood tests, and X-rays, if medically indicated. Visits may be more frequent, if necessary.

ELIGIBILITY:
* INCLUSION CRITERIA:

Diagnosis of HCV-CV: must have all of the following

HCV infection documented by serology and/or plasma HCV RNA.

One or more organ system with objective evidence of active vasculitis such as:

Palpable purpura;

Glomerulonephritis (defined by the presence of glomerular hematuria and/or new or worsening proteinuria);

Acute peripheral neuropathy.

Detectable cryoglobulins and/or RF.

Failure of treatment with IFN-alpha and ribavirin to control manifestations of HCV-CV OR intolerance to IFN-alpha/ribavirin regimen.

Patients must have a personal physician responsible for the care of their HCV.

Ages of 18 and 75 years

Willingness to use effective contraception during and for 12 months following Rituximab treatment. Effective contraception methods include abstinence, surgical sterilization of either partner, barrier methods such as diaphragm, condom, cap or sponge, or hormonal contraception.

EXCLUSION CRITERIA:

Recent (within 4 weeks) initiation of or increase in immunosuppressive therapy.

Active systemic infection (other than hepatitis C).

Pregnancy or breast feeding.

Prior treatment with Rituximab.

Known allergy to murine proteins.

Significant renal insufficiency (creatinine clearance less than 30 ml/min).

Presence of life-threatening HCV-CV; defined as rapidly progressive glomerulonephritis (defined as a doubling of the serum creatinine over a 3 month period), CNS vasculitis, cardiac disease due to active vasculitis, or GI vasculitis (defined by ischemic bowel, perforation, or infarction).

Significant hepatic insufficiency as manifested by Child-Pugh classification of B or C.

History of variceal bleeding, encephalopathy.

History of liver transplantation.

Co-infection with either HBV or HIV.

Any underlying medical condition that in the judgment of the investigator would put the patient at increased risk for serious infusion-related adverse events.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2001-12; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Sneller, MD, Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ferri C, Greco F, Longombardo G, Palla P, Moretti A, Marzo E, Fosella PV, Pasero G, Bombardieri S. Antibodies to hepatitis C virus in patients with mixed cryoglobulinemia. Arthritis Rheum. 1991 Dec;34(12):1606-10. doi: 10.1002/art.1780341221. PMID 1660716
- [Background] Misiani R, Bellavita P, Fenili D, Borelli G, Marchesi D, Massazza M, Vendramin G, Comotti B, Tanzi E, Scudeller G, et al. Hepatitis C virus infection in patients with essential mixed cryoglobulinemia. Ann Intern Med. 1992 Oct 1;117(7):573-7. doi: 10.7326/0003-4819-117-7-573. PMID 1326246
- [Background] Cacoub P, Fabiani FL, Musset L, Perrin M, Frangeul L, Leger JM, Huraux JM, Piette JC, Godeau P. Mixed cryoglobulinemia and hepatitis C virus. Am J Med. 1994 Feb;96(2):124-32. doi: 10.1016/0002-9343(94)90132-5. PMID 7509124
- [Derived] Sneller MC, Hu Z, Langford CA. A randomized controlled trial of rituximab following failure of antiviral therapy for hepatitis C virus-associated cryoglobulinemic vasculitis. Arthritis Rheum. 2012 Mar;64(3):835-42. doi: 10.1002/art.34322. PMID 22147444

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between June 2002 and April 2010, a total of 24 patients were enrolled in the study. Twelve patients randomized to the rituximab group and 12 patients to the control group.
Pre-assignment Details: A total of 47 patients were screened for randomization into this study. Eighteen patients did not meet one or more of the above eligibility criteria. Five eligible patients elected not to enroll in the study because of concerns about potential rituximab toxicity. The remaining 24 patients were enrolled in the study and underwent randomization
Groups:
- Immediate Treatment: Patients receive treatment with four weekly infusions of rituximab immediately following randomization.
- Standard Therapy: Receives standard therapy. After 6 months, they are eligibile to cross over and receive four weekly infusions of rituximab.
Period: Overall Study
Arm/Group | Immediate Treatment | Standard Therapy
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Treatment | Standard Therapy | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 52 (5.6) | 51 (4) | 51 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 10 | 8 | 18
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients in Remission
Description: The primary endpoint was the difference in rate of remission between the 2 arms at 6 months from study entry.
Time Frame: month 6
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Immediate Treatment | Standard Therapy
Number analyzed (Participants) | 12 | 12
percent of participants | 83 [52 to 98] | 8 [2 to 38]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Only adverse events that were grade 3 or greater and were possibly or probably related to the study drug were collected and analyzed for the purposes of this study
Arm/Group | Immediate Treatment | Standard Therapy
Serious Adverse Events (participants affected / at risk) | 6/12 | 8/12
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Treatment (N=12) | Standard Therapy (N=12)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
AST elevation > grade 3 (Hepatobiliary disorders) | 3 (4) | 3 (3)
Infection (Infections and infestations) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
The study was not blinded. In addition, the study was limited to patients who had failed antiviral therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes